CLINICAL TRIAL: NCT01629524
Title: Influence of Tumor Associated Immunity on the Number of Lymph Node Retrieved After Colorectal Cancer Surgery (Preliminary Study)
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-08
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and postoperative specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Colorectal cancer patients undergoing elective colorectal resection

SUMMARY:
Hypothesis of this study is that increased immunity of primary tumor affects the increased number of lymph node retrieved. This study investigates whether immunity-related cytokine expression on primary tumor, colonic mucosa, and serum is associated with the number of lymph node retrieved in colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed colorectal cancer 2. Non-metastatic cancer (cTNM I, II, or III) 3. Over 20 years of age 4. Curative resection (R0)

Exclusion Criteria:

* 1. Patient with distant metastasis 2. History of chemotherapy or radiation therapy for malignancy 3. Patient receiving immunosuppressive or anti-inflammatory treatment 4. Hereditory colorectal cancer 5. Preoperative chemoradiation therapy for colorectal cancer 6. Pregnancy 7. Emergency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients diagnosed with clinically TNM I, II, or III stage
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Association between immune related cytokine and number of lymph nodes retrieved. | 2 months after surgery
  Immunity related cytokine - IL-12, IFN-r, GM-CSF, IL-4, TNF-a, IL-6, IL-8, IL-10, TGF-b1, CXCR4, SDF1, HGF, VEGF - expression is assessed using Bioplex assay. Patient serum is taken one day before surgery. Primary tumor and colonic mucosal tissue are taken just after surgery. Bioplex assay is performed after patients' enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Wonji Christian Hospital, Wŏnju, South Korea

REFERENCES:
- [Derived] Kim YW, Kim SK, Kim CS, Kim IY, Cho MY, Kim NK. Association of serum and intratumoral cytokine profiles with tumor stage and neutrophil lymphocyte ratio in colorectal cancer. Anticancer Res. 2014 Jul;34(7):3481-7. PMID 24982357